CLINICAL TRIAL: NCT04164225
Title: Identifying Brain Mechanisms Related to Body Awareness Using QiGong to Relieve Chronic Low Back Pain
Brief Title: Feasibility of Identifying Brain Mechanisms of Qigong and Behavioral Outcomes After Qigong Practice in People With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PMR-2019-27351
Record Dates: First submitted 2019-04-24; First posted 2019-11-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong (Experimental): Qigong exercises, focused on a mind-body connection
  Interventions: Behavioral: Qigong Exercise
- P.Volve (Active Comparator): P.Volve exercises, focused on just physical movement
  Interventions: Behavioral: P.Volve Exercises

INTERVENTIONS:
Behavioral: Qigong Exercise — Participants with chronic low back pain will follow the free "5 elements Qigong healing class" (estimate of 6 hours) at the Spring Forest Qigong center and then practice the "5 elements healing Qigong" at home 3 times a week for 40 minutes with a freely available online video, for 12 weeks. A weekly group session (1 hour) will be conducted at the Brain Body Mind Lab with the principal investigator to address questions and demonstrate movements if needed.
  Arms: Qigong
Behavioral: P.Volve Exercises — P.Volve exercise focuses on low impact core strengthening, core stabilization, and stretching. The program is similar in delivery as Qigong (i.e., online videos). An introductory class (estimate of 2.5h) will be given by the P.Volve team, the principal investigator, and a physical therapist who has experience with P.Volve exercises. Participants will access online videos for individual home practice in 40min/session, 3x/week for 12 weeks. Participants will receive a P.ball for some exercises, while other exercises are done with no equipment. Tailored videos will be available for those with cLBP. A weekly group session (1 hour) will be conducted at the Brain Body Mind Lab with the principal investigator to address questions and demonstrate movements if needed.
  Arms: P.Volve

SUMMARY:
The long-term objective of this investigation is to identify how Qigong affects brain function in brain areas relevant to patients with chronic low back pain (cLBP), thereby setting a foundation from which to perform further clinical research.

DETAILED DESCRIPTION:
The central hypothesis of this investigation is that, in adults with cLBP, practicing Qigong compared to exercise will result in reduced pain and improved body awareness and proprioception (primary behavioral endpoints), disability, balance, core muscle strength, and other CLBP symptoms will be secondary behavioral endpoints.To test this hypothesis, the investigators will assess (1) participant recruitment and retention ; (2) adherence to interventions, engagement/satisfaction with the program; and (3) changes in body awareness-related brain activation and connectivity pre-post intervention (Qigong vs exercise) related to primary endpoints of pain perception, body awareness and objective measures of lower limb proprioception.

ELIGIBILITY:
Inclusion Criteria:

- Adults with chronic low back pain

Exclusion Criteria:

* Those with cognitive problems
* Those unable to speak or understand instructions
* Those who have nerve problems, fractures, or infections
* Those who do not speak English
* Those with severe deficit in motor imagery or in vision (both are used in MRI tasks)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Numeric Rating Scale (NRS) | baseline, 15 weeks
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. Pain is rated on a scale of 0-10, with higher scores indicating greater pain intensity.
Change in Revised Body Awareness Rating Questionnaire (BARQ) | baseline, 15 weeks
  The Body Awareness Rating Questionnaire (BARQ) is a self-report questionnaire designed to capture how individuals with long-lasting musculoskeletal pain reflect on their own body awareness. This questionnaire contains 12 items rated on a scale from 0 (completely disagree) to 3 (completely agree). The total score is a sum of all items. Lower scores indicate greater body awareness.
Change in Mindfulness Attention Awareness Scale (MAAS) | baseline, 15 weeks
  The MAAS is a 15-item scale designed to assess a core characteristic of mindfulness. Items are rated on a scale from 1 (almost always) to 6 (almost never). The total score is an unweighted mean of the 15 item scores.
Change in Five-Facet Mindfulness Questionnaire (FFMQ) | baseline, 15 weeks
  The FFMQ is a 39-item scale measuring five facets of mindfulness: observing (items 1, 6, 11, 15, 20, 26, 31, and 36), describing (items 2, 7, 12R, 16R, 22R, 27, 32, and 37), acting with awareness (items 5R, 8R, 13R, 18R, 23R, 28R, 34R, 38R), non-judging of inner experience (items 3R, 10R, 14R, 17R, 25R, 30R, 35R, 39R), and non-reactivity to inner experience (items 4, 9, 19, 21, 24, 33). Items are rated on a scale from 1 (never or very rarely true) to 5 (very often or always true). Items marked with "R" are scored in reverse. Sub scale and total scale scores can be calculated by sum or unweighted mean. Higher scores indicate higher levels of mindfulness.
Change in Proprioception | baseline, 15 weeks
  Lower-limb proprioception will be measured by a lower limb device that produces assessment of proprioceptive acuity and sensitivity of the ankle and/or knee joint in the sagittal plane. Output is measured in degrees of joint motion of the ankle and knee.
Change in Postural Awareness Scale (PAS) | baseline, 15 weeks
  The PAS is a 12-item scale, which was developed in order to measure self-reported awareness of body posture in patients with chronic pain and to evaluate potential changes in postural awareness induced by a multimodal mind-body training program. Item responses range from 1 (not at all true about me) to 7 (very true about me). Six items are reversely scored, so that higher score values consistently indicate higher postural awareness. Total scores are a sum of items scores and range from 13 to 91, with higher scores indicating greater postural awareness

SECONDARY OUTCOMES:
Change in Modified Roland Morris Disability Questionnaire | baseline, 15 weeks
  The Modified Roland Morris Disability Questionnaire, designed to assess self-rated physical disability caused by low back pain, contains 23 items. Items are scored 0 (no) or 1 (yes). Total scores are calculated as a sum with higher scores indicated greater physical disability caused by low back pain.
Change in Fear-Avoidance Beliefs Questionnaire (FABQ) | baseline, 15 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ), a patient-reported questionnaire focusing on how a patient's fear of physical activity and work may affect their low back pain and disability, contains 16 items rated on a 7-point Likert from 0 (completely disagree) to 6 (completely agree). Total scores are calculated as a sum with a maximum score of 96. Higher scores indicated more strongly-hold fear avoidance beliefs.
Change in Pain Self-Efficacy questionnaire (PSEQ) | baseline, 15 weeks
  The Pain Self-Efficacy questionnaire (PSEQ) is a 10-item questionnaire measuring a patient's confidence in their ability to complete a task despite pain. Items are rated on a scale from 0 (not at all confident) to 6 (completely confident). Total scores are a sum of the 10 items scores with a maximum score of 60. Lower scores indicate greater pain-related disability.
Change in Tampa Scale for Kinesiophobia | baseline, 15 weeks
  The Tampa Scale for Kinesiophobia is a 17-item questionnaire measuring fear related to exercise and movement. Items are rated on a scale of 1 (strongly disagree) to 4 (strongly agree). A total score is calculated by summing the individual item scores after inversion of the individual scores for items 4, 8, 12 and 16. Higher scores indicated greater kinesiophobia.
Change in Core Muscle Stabilization - Prone | baseline, 15 weeks
  Participants are asked to perform a prone bridge position. The length of time the position is held is recorded in seconds.
Change in Core Muscle Stabilization - Supine | baseline, 15 weeks
  Participants are asked to perform a supine bridge position. The length of time the position is held is recorded in seconds.
Change in Balance Test - Right Leg | baseline, 15 weeks
  Participants are asked to stand on one leg. The length of time the position is held is recorded in seconds.
Change in Balance Test - Left Leg | baseline, 15 weeks
  Participants are asked to stand on one leg. The length of time the position is held is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, PhD,MSPT,PT, Principal Investigator — University of Minnesota
Locations (1):
- Children's Rehabilitation Center, 426 Church Street SE Room 302 - Brain Body Mind Lab Minneapolis, MN 55455, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Van de Winckel A, Zhang L, Hendrickson T, Lim KO, Mueller BA, Philippus A, Monden KR, Oh J, Huang Q, Sertic JVL, Ruen J, Konczak J, Evans R, Bronfort G. Identifying body awareness-related brain network changes after Spring Forest Qigong practice or P.Volve low-intensity exercise in adults with chronic low back pain: a feasibility Phase I Randomized Clinical Trial. medRxiv [Preprint]. 2023 Mar 1:2023.02.11.23285808. doi: 10.1101/2023.02.11.23285808. PMID 36824785
- See also: Evaluating the effect and mechanism of Qigong in people with chronic low back pain — https://www.med.umn.edu/rehabmedicine/research/identifying-qigong-brain-changes